CLINICAL TRIAL: NCT07038460
Title: A Multicenter Phase II Randomized Trial of Limertinib Followed by Sintilimab and Chemotherapy vs. Limertinib Followed by Limertinib and Chemotherapy as Neoadjuvant Therapy in Resectable Stage II-IIIB EGFR-Mutant NSCLC
Acronym: NEO-LISI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wen-zhao ZHONG (Other)
Responsible Party: Sponsor-Investigator, Wen-zhao ZHONG, Ph.D, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangdongPPHosp
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Resectable Non-small Cell Lung Cancer
Keywords: NSCLC; EGFRmut; Limertinib; Sintilimab
MeSH Terms: interventions — Surgical Procedures, Operative; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: Limertinib+sintilimab+chemotherapy; Procedure: surgery; Drug: Osimertinib
- Control Group (Active Comparator)
  Interventions: Drug: Limertinib+chemotherapy; Procedure: surgery; Drug: Osimertinib

INTERVENTIONS:
Drug: Limertinib+sintilimab+chemotherapy — Experimental group patients receive Limertinib for 6 weeks. Within 7 days thereafter, imaging assessment will be performed. If no progression is observed, experimental group patients discontinue therapy for 1 week, then receive Sintilimab + Carboplatin/Cisplatin + Pemetrexed every 3 weeks for 3 cycles.
  Arms: Experimental Group
Drug: Limertinib+chemotherapy — Control group group patients receive Limertinib for 6 weeks. Within 7 days thereafter, imaging assessment will be performed. If no progression is observed, control group patients receive Lilotinib for next 9 weeks + Carboplatin/Cisplatin + Pemetrexed every 3 weeks for 3 cycles.
  Arms: Control Group
Procedure: surgery — The surgical procedure may involve minimally invasive surgery (video-assisted thoracoscopic surgery, robot-assisted surgery) or open thoracotomy. The surgical methods include lobectomy, combined lobectomy, pneumonectomy, sleeve resection, and ipsilateral systematic mediastinal lymph node dissection (for left-sided tumors, stations 4L, 5, 6, 7, and 9 should be included; for right-sided tumors, at least stations 2R, 3A, 4R, 7, and 9 should be included).
Drug: Osimertinib — Adjuvant treatment with Osimertinib for 2 years

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of neoadjuvant therapy with Limertinib Followed by Sintilimab and Chemotherapy in resectable Stage II-IIIB EGFR-Mutant NSCLC. Untreated stage II-IIIB NSCLC (AJCC 8th edition) patients assessed as surgically resectable by investigators will be randomized 1:1 into the experimental or control group after signing informed consent and meeting eligibility criteria. All patients receive Limertinib for 6 weeks. Within 7 days thereafter, imaging assessment will be performed. If no progression is observed, experimental group patients discontinue therapy for 1 week, then receive Sintilimab + Carboplatin/Cisplatin + Pemetrexed every 3 weeks for 3 cycles; control group patients receive Limertinib for 9 weeks and Carboplatin/Cisplatin + Pemetrexed every 3 weeks for 3 cycles. Preoperative tumor assessment is required. Surgery will be performed 2-6 weeks (±7 days) after the first dose of the final cycle. Then patients will recieve 2-year adjuvant Osimertinib starting 1 month post-surgery. If imaging assessment after 6 weeks of limertinib treatment shows lesion enlargement but remains confined to stage II-IIIB, the investigator will decide whether the patient continues study treatment or not; if progression occurs to unresectable stage III or advanced disease, the patient must discontinue. The primary endpoint is pathological complete response (pCR) rate.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form
2. Age: 18-75 years.
3. Cytologically/histologically confirmed (via percutaneous lung puncture, bronchoscopy, mediastinoscopy, etc.), previously untreated stage II-IIIB (IASLC 8th Edition Thoracic Tumor Classification) lung adenocarcinoma.
4. Tumor tissue or blood samples confirmed as EGFR-sensitive or rare mutation-positive by laboratory testing
5. Must provide archived tumor tissue or newly resected tumor biopsy samples for PD-L1 IHC testing during screening.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
7. Measurable lesions per RECIST v1.1.
8. Surgically evaluated as eligible for local surgical resection (adequate pulmonary/organ function).Surgically evaluated as eligible for local surgical resection (adequate pulmonary/organ function).
9. Adequate organ and bone marrow function (within 7 days prior to enrollment; no corrective therapies within 14 days prior to testing): • Hematology: ANC ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥100 g/L. • Hepatic: Total bilirubin ≤1.5×ULN; AST/ALT ≤2.5×ULN; albumin ≥35 g/L. • Renal: Serum creatinine ≤1.5×ULN; CrCl ≥60 mL/min (Cockcroft-Gault formula); urine protein <2+ or 24-hour urine protein <1 g. Cockcroft-Gault formula: • Female: CrCl = [(140 - age) × weight (kg) × 0.85] / [72 × serum creatinine (mg/dL)]. • Male: CrCl = [(140 - age) × weight (kg)] / [72 × serum creatinine (mg/dL)]. • Coagulation: INR ≤1.5×ULN; PT/APTT ≤1.5×ULN.
10. For women of childbearing potential: Negative urine/serum pregnancy test within 7 days prior to first dose. Confirmatory blood test required if urine test is positive.

Exclusion Criteria:

1. Patients with stage I or IV NSCLC who have previously received systemic anti-tumor therapies (e.g., ICIs, targeted therapy, chemotherapy).
2. Active known or suspected autoimmune diseases (exceptions: type I diabetes, hypothyroidism requiring hormone replacement only, non-progressive skin conditions like vitiligo/psoriasis/alopecia).
3. Active hepatitis B (HBsAg-positive) or hepatitis C (HCV RNA-positive). Patients with resolved HBV infection (HBsAg-negative, HBcAb-positive) must provide HBV DNA-negative results. HCV antibody-positive patients require negative HCV RNA PCR.
4. HIV-positive or AIDS history.
5. Arterial thrombosis within 6 months, or deep vein thrombosis/pulmonary embolism within 3 months.
6. Uncontrolled angina, arrhythmias, or congestive heart failure.
7. Active malignancies within 5 years (except cured cervical/cutaneous carcinoma in situ, superficial bladder/prostate/breast cancer).
8. Contraindications to local therapies (surgery, radiotherapy, or intervention) per investigator judgment.
9. Hypersensitivity to sintilimab, limertinib, chemotherapy agents, or excipients.
10. Unwillingness to sign informed consent or comply with follow-up.
11. Any condition compromising trial integrity or patient safety, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | Up to approximately 6 weeks following completion of surgery
  Pathology evaluation confirmed no residual tumor cells in the resected specimen and regional lymph nodes.

SECONDARY OUTCOMES:
Major Pathological Response (mPR) Rat | Up to approximately 6 weeks following completion of surgery
  mPR rate is defined as ≤ 10% residual invasive viable tumor in both the primary tumor (lung) and the sampled lymph nodes after neoadjuvant therapy.
Event Free Survival (EFS) | Up to approximately 2.5 years following the beginning of Post-operative Assessment baseline
  EFS is defined as the time from randomization to the first recorded time to any first documented progression, recurrence or death, which occurs first.
Disease free survival (DFS) | Up to approximately 2 years following the begining of Post-operative Assessment baseline
  DFS is defined as the time from surgery to disease recurrence or death due to any cause.
Overall survival (OS) | Up to approximately 2.5 years
  OS is defined as the time from randomization to death due to any cause.
Objective response rate(ORR) | Up to approximately 2 weeks before surgery
  The proportion of patients in whom tumor volume reduction reached the predetermined criteria and was maintained for the minimum required duration is the sum of the complete response (CR) and partial response (PR) rates.
Safety parameters:AE | Up to approximately 2.5 years
  The relationship of study drug and the severity of all adverse events (AEs), treatment emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), immune-related adverse events (irAEs), serious adverse events (SAEs), infusion-related reactions (IRRs) and surgery delay rate.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical Univercity, Guangzhou, Guangdong
  - Guangdong Province People's Hospital, Guangzhou, Guangdong
  - Sun Yet-Sen University Cancer Center, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang